CLINICAL TRIAL: NCT01703598
Title: Clinical Outcomes of Deep Brain Stimulator Electrodes Placed Using Intraoperative Computed Tomography and Frameless Stereotaxis Versus Microelectrode Recording and Frame-based Stereotaxis
Brief Title: Clinical Outcomes of Deep Brain Stimulator (DBS) Electrodes Placed Using Intraoperative Computed Tomography (CT) and Frameless Stereotaxis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Matthew Brodsky, Principal Investigator, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00007508
Record Dates: First submitted 2011-09-09; First posted 2012-10-10 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: Asleep Deep Brain Stimulation
Oversight: Data Monitoring Committee: No

ARMS (1):
- DBS surgery (Experimental): Single arm
  Interventions: Device: Deep Brain Stimulation; Procedure: DBS surgery

INTERVENTIONS:
Device: Deep Brain Stimulation — Placement of Deep Brain Stimulation electrodes
Procedure: DBS surgery — Placement of DBS electrodes

SUMMARY:
The purpose of this study is to determine whether performing deep brain stimulation surgery for Parkinson's disease using intraoperative imaging and frameless stereotaxis is noninferior to using frame-based stereotaxy and microelectrode recording.

DETAILED DESCRIPTION:
Background: Frame-based stereotaxis and microelectrode recording (MER) with mapping of target structures has been the gold standard for deep brain stimulator (DBS) implantation. Though supported by historical considerations, no Class I or II evidence exists that MER adds significant value to the DBS implant procedure. With the advent of advanced magnetic resonance imaging (MRI) and computed tomography (CT) imaging, particularly intra-operative imaging, the argument for the continued use of MER during DBS implantation has been substantially weakened. One rationale for pursuing CT-guided intraoperative imaging is due to presumed increase in patient comfort with this method. DBS implantation with MER requires that the patient remain awake during the entire procedure. , MER with frame-based stereotaxis requires the patient to keep their head in a fixed position for a prolonged period of time during which time they remain awake, causing significant patient discomfort. Furthermore, Parkinson's disease patients must withhold their PD meds for a minimum of 12 hours prior to the procedure adding a sometimes significant degree of discomfort and anxiety to the procedure.

Objective: The goal of this study is to compare the clinical outcomes of DBS electrodes placed using intraoperative CT and frameless stereotaxis with those placed using MER and frame-based stereotaxis.

Design: The proposed study will be a prospective non-interventional data collection study.

Setting and Subjects: Subjects for this study will be idiopathic Parkinson's disease patients identified from the Oregon Health & Science University movement disorder clinic as candidates for deep brain stimulation therapy. Enrollment will continue until fifty subjects have been implanted with electrodes using frameless stereotaxis and intraoperative CT. Data regarding quality of life, motor control, and amount of time during the day without levodopa side effects will be collected pre-operatively and post-operatively. This data will be compared to historical controls who have been implanted with DBS electrodes using MER and frame-based stereotaxis. All surgical procedures will involve only Federal Drug Administration (FDA) approved stereotactic equipment, used in the manner for which they have been approved. All clinic procedures are standard of care for movement disorders patients in the deep brain stimulation program.

Intervention: This study will be a non-interventional data collection study.

Measurements: Data regarding patient age, diagnosis, intracranial target, complications, Unified Parkinson's Disease Rating Scale UPDRS Parts 3 (motor examination) and 4 (drug side effects), Parkinson's Disease Quality of life PDQ-39, 3 day motor diary, 3 month falls diary, neuropsychiatric evaluation and days in hospital following surgery will be collected.

Analysis: The patients will be examined prior to DBS placement both on and off dopaminergic medications. They will then be examined 3 months and 6 months following DBS placement both on and off drug with stimulator on after programming parameters have been optimized. The following measures will be performed:

* Change in UPDRS Parts 3 and 4
* Change in PDQ-39
* Change in amount of time patient is experiencing Parkinson's disease symptoms and/or side effects of treatment.
* Change in number of falls
* Change in neuropsychiatric evaluation, including:
* Beck Depression Inventory-II (BDI-II)
* Mattis Dementia Rating Scale-Second Edition (DRS-2)
* Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)
* Symptom Checklist-90-Revised (SCL-90-R)
* Wechsler Abbreviated Scale of Intelligence (WASI) We will also compare the number of days spent in hospital following surgery. Adverse events related to the surgery will be captured.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease patients identified by OHSU movement disorders neurologists as deep brain stimulation surgical candidates

Exclusion Criteria:

* Subjects who have already undergone implantation of DBS electrodes 2.Age < - - 18 years
* Surgical target site other than subthalamic nucleus or globus pallidus pars interna
* Subjects who choose to undergo MER and frame-based stereotaxis for the placement of electrodes.
* Patients who will receive follow up neurology care and DBS programming at centers other than OHSU.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brodsky, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Derived] Brodsky MA, Anderson S, Murchison C, Seier M, Wilhelm J, Vederman A, Burchiel KJ. Clinical outcomes of asleep vs awake deep brain stimulation for Parkinson disease. Neurology. 2017 Nov 7;89(19):1944-1950. doi: 10.1212/WNL.0000000000004630. Epub 2017 Oct 6. PMID 28986415

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | DBS Surgery
Started | 69
Completed | 69
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: The analysis population is the same as the baseline population
Arm/Group | DBS Surgery
Number analyzed (Participants) | 69
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.1 (7.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 46
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Motor OFF Ldopa UPDRS
Description: Change in motor UPDRS in OFF Levodopa state. The range of this outcome is from 0 to 108, a higher number indicated a worse clinical state.
  The number represents units on this scale.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: motor UPDRS
Arm/Group | DBS Surgery
Number analyzed (Participants) | 69
motor UPDRS | 14.8 (8.9)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | DBS Surgery
All-Cause Mortality (participants affected / at risk) | 0/69
Serious Adverse Events (participants affected / at risk) | 0/69
Other Adverse Events (participants affected / at risk) | 0/69

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-06): https://cdn.clinicaltrials.gov/large-docs/98/NCT01703598/Prot_SAP_000.pdf